CLINICAL TRIAL: NCT06040619
Title: Implementation of Therapy Together With the State of Texas Early Childhood Intervention Program
Brief Title: Implementation of Therapy Together
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Angela Shierk, Clinical Scientist, Texas Scottish Rite Hospital for Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0553
Record Dates: First submitted 2023-08-28; First posted 2023-09-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: constraint induced movement therapy; caregiver coaching
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Pilot randomized control trial comparing treatment group to usual care. The usual care group will have the option to cross over to the treatment group after 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy Together (Experimental): Participants will complete the 8-week Therapy Together program.
  Interventions: Behavioral: Therapy Together
- Usual Care (Active Comparator): Participants will complete 8 weeks of usual care in early intervention.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Therapy Together — 8-week caregiver-led pediatric constraint-induced movement therapy program
  Arms: Therapy Together
Behavioral: Usual Care — 8 weeks of usual care received in an early intervention therapy program
  Arms: Usual Care

SUMMARY:
The goal of this clinical trial is to learn about the implementation of Therapy Together, a pediatric constraint-induced movement therapy program in young children with unilateral cerebral palsy. The main question[s] it aims to answer are:

* Is the Therapy Together program effective in improving hand function and occupational performance compared to usual care?
* Is it feasible to implement the Therapy Together program within the standard care, early intervention framework?

Participants will participate in an 8-week pediatric constraint-induced movement therapy program. Researchers will compare the group completing the Therapy Together Program to a group that is receiving usual care to see if there is a difference in the change in hand function, occupational performance, and development.

DETAILED DESCRIPTION:
A randomized waitlist control trial with early intervention therapists, infants/toddlers (ages 3 mo - 5 yrs 11 mo) with unilateral cerebral palsy (or at risk for developing cerebral palsy) and caregivers comparing Therapy Together to usual care followed by semi-structured interviews with caregivers and therapists will be utilized to examine the implementation and effectiveness of Therapy Together within early intervention.

Therapy Together Program:

The Therapy Together program includes caregiver education and coaching on implementing therapeutic activities that are play-based, age-appropriate, and tailored to meet goals to improve arm/hand function. The child and caregiver complete 8 sessions with their therapist. The therapist is trained to educate the caregiver on the Therapy Together program, demonstrate how to engage the child in therapeutic activities, and observe the caregiver implement the program during each weekly session. The first 7 intervention visits focus on constraint-induced movement therapy (CIMT) and the final intervention visit focuses on bimanual therapy (use of two hands).

ELIGIBILITY:
Inclusion Criteria:

* at risk for developing cerebral palsy or have been diagnosed with cerebral palsy
* children ages 3 months to 5 years 11 months
* present with asymmetric hand use
* present with a unilateral upper limb impairment
* able to visually attend to objects
* demonstrate an interest in objects
* attempt to reach for or grasp objects with the impaired upper extremity

Exclusion Criteria:

* uncontrolled epilepsy
* significant visual impairment
* severe behavioral problems
* inability to complete the assessment protocol.

Ages: 3 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mini-Assisting Hand Assessment | baseline, pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Mini-Assisting Hand Assessment is an observation-based, criterion-referenced assessment that assesses bimanual hand function for children with cerebral palsy aged 8-18 months (measured in logits/units)
Assisting Hand Assessment | baseline, pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Assisting Hand Assessment is an observation-based, criterion-referenced assessment that assess bimanual hand function for children with cerebral palsy, aged 18 months-12 years (measured in logits/units)
Hand Assessment for Infants | baseline, pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Hand Assessment for Infants is an observation-based, criterion-referenced and norm-referenced assessment of unilateral and bimanual hand function for children with cerebral palsy aged 3 months-12 months (measured in logits/units)

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | baseline, pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Canadian Occupational Performance Measure is an interview-based assessment of self-perception of performance of everyday living activities (measured on a scale from 1-10)
Developmental Assessment for Young Children, Second Edition (DAYC-2) | baseline, pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Developmental Assessment for Young Children is an interview and observation based norm-referenced developmental assessment (raw scores 0 or 1, converted to standard scores)
Measure of Hand and Arm Performance | baseline, pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Measure of Hand and Arm Performance is a criterion-referenced, observational assessment of hand and arm use based on observation, measured on a scale of 1-10

OTHER OUTCOMES:
Pre-training and Post-training Therapist Survey | Baseline, pre-intervention and within 1 month of post-intervention
  The pre-training and post-training survey includes questions on knowledge, appropriateness, and acceptability of pediatric constraint-induced movement therapy (includes likert scale questions, demographic questions, and open ended qualitative responses)
Interviews with therapists and caregivers | Within 1 month of post intervention
  Interviews to explore feasibility, fidelity, cost, appropriateness, and acceptability, qualitative data
Weekly Caregiver Log | weekly for 8 weeks
  The caregiver log includes feasibility (time), stress, and impact on unilateral and bimanual hand function measured using a likert scale of 1-4
Weekly Therapist Log | weekly for 8 weeks
  Weekly therapist logs include feasibility, fidelity, cost of the program, measured using a checklist, and qualitative responses

CONTACTS AND LOCATIONS:
Overall Officials: Angela Shierk, PhD, Principal Investigator — Scottish Rite for Children
Locations (1):
- Scottish Rite for Children, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No